CLINICAL TRIAL: NCT01032161
Title: Perioperative Risk Factors for Postoperative Delirium in Children Following General Anesthesia
Brief Title: Perioperative Risk Factors for Postoperative Delirium in Children
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Other Study IDs: TIHMZK02002
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Delirium, Postoperative
Keywords: Delirium; Postoperative; Non-cardiovascular surgery; Post-anaesthesia care unit; patients between 3 to 12 years old; undergoing selective non-cardiac surgery; under general anesthesia; surgery; general anesthesia
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Delirium: Delirium was determined by RASS-PAEDS
- no Delirium: no Delirium was determined by RASS-PAEDS

SUMMARY:
Despite recent advances in postoperative delirium research, the proportion of children with postoperative delirium is still high. Although postoperative delirium is a frequent complication and is associated with the need for more inpatient hospital care and longer length of hospital stay, little is known about risk factors for recovery room delirium (RRD) occurred in postanaesthesia care unit. The aim of the study was to determine pre- and intraoperative risk factors for the development of RRD among children undergoing non cardiovascular surgery.

DETAILED DESCRIPTION:
Recovery room delirium (RRD) defined as delirium occurred in PACU was diagnosed according to RASS-PAEDS criteria. Pre-, intra-, and postoperative data of patients undergoing elective non cardiovascular surgery were prospectively collected, univariate and multivariate logistic regression were performed to find the risk factors related to postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* between 3 to 12 years old
* elective non-cardiovascular surgery
* general anesthesia

Exclusion Criteria:

* under regional anaesthesia
* instable vital sign
* without consent form
* underwent neurosurgery
* history of primary neurologic diseases
* stayed less than 10min in PACU
* received general anaesthesia but recovered in locations outside the recovery room

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients between 3 to 12 years old, who were admitted to the PACU after elective non-cardiac surgery under general anaesthesia during regular working hours (9:00Am to 5:00Pm)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The presence of delirium in post anesthesia care unit (PACU) and in ward determined by RASS-PAEDS criteria | at 1, 8, 16, 24, 48 and 72 postoperative hour

SECONDARY OUTCOMES:
Maximal and minimal heart rate in PACU | every 15 min during PACU stay
Pulse Oximeter Oxygen Saturation (SpO2) in PACU | every 15 min during PACU stay
Hospital-length of stay | before discharge
Total health care fees | during hospital stay
Quality of recovery measured by PACBIS criteria | at 1, 8, 16, 24, 48 and 72 postoperative hour

CONTACTS AND LOCATIONS:
Overall Officials: Chuanhan Zhang, M.D., Study Director — Department of Anaesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology; Yuke Tian, M.D., Study Chair — Department of Anaesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China